CLINICAL TRIAL: NCT01904253
Title: An Open-Label, Randomized, Phase 2 Study Comparing TAS-102 Versus Topotecan or Amrubicin in Patients Requiring Second-Line Chemotherapy for Small Cell Lung Cancer That is Refractory or Sensitive to First-Line Platinum-Based Chemotherapy
Brief Title: A Phase 2 Study Comparing TAS-102 Versus Topotecan or Amrubicin to Treat Small Cell Lung Cancer Following Platinum-Based Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The preliminary data does not suggest any safety signal, but an ad hoc interim analysis showed an imbalance of PFS between the two arms
Sponsor: Taiho Oncology, Inc. (Industry)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPU-TAS-102-201; 2012-004793-26 (EudraCT Number)
Record Dates: First submitted 2013-07-12; First posted 2013-07-22 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: Second line Small Cell Lung Cancer, (SCLC), Refractory or Sensitive to First line Platinum based chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — trifluridine tipiracil drug combination; amrubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAS-102 (Experimental)
  Interventions: Drug: TAS-102
- Investigator Choice of Amrubicin or Topotecan (Active Comparator): Investigator Choice of Amrubicin (Japan only) or Topotecan (Europe and Japan)
  Interventions: Drug: Amrubicin (Japan); Drug: Topotecan (Japan/Europe)

INTERVENTIONS:
Drug: TAS-102 — 35 mg/m2/dose, orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Arms: TAS-102
Drug: Amrubicin (Japan) — Patients will receive treatment administered according to the country-specific approved prescribing information
  Other Names: Calsed
  Arms: Investigator Choice of Amrubicin or Topotecan
Drug: Topotecan (Japan/Europe) — Patients will receive treatment administered according to the country-specific approved prescribing information
  Other Names: Hycamptin; Hycamtin
  Arms: Investigator Choice of Amrubicin or Topotecan

SUMMARY:
The purpose of this trial is to compare the effects of TAS-102 with either amrubicin or topotecan (drugs used in Small Cell Lung Cancer) on lung cancer to find out the effects on survival, how much time may pass without disease progression, and the safety of TAS-102.

DETAILED DESCRIPTION:
This is a multicenter, open-label, two-arm, randomized Phase 2 study of TAS-102 versus Investigator's choice of therapy in patients requiring second-line chemotherapy for SCLC refractory or sensitive to first-line platinum-based chemotherapy. Investigator's choice of therapy is defined as second-line chemotherapy with IV topotecan (Europe/Japan) or IV amrubicin (Japan). Patients will be stratified by response to first-line platinum-based chemotherapy (sensitive vs refractory). Sensitive patients are defined as patients who did not progress within 90 days after the last dose, and refractory patients are defined as patients who never responded or who responded but had radiologic progression < 90 days after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Is ≥18 years of age for patients enrolled in Europe; or ≥20 years of age for patients enrolled in Japan
3. Has definitive histologically or cytologically confirmed SCLC (limited or extensive disease)
4. Has progressed or had recurrence within 30 days prior to randomization
5. Has at least one measurable lesion, as defined by RECIST criteria version 1.1
6. ECOG performance status of 0, 1, or 2
7. Is able to take medications orally
8. Has adequate organ function (bone marrow, kidney and liver)
9. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Has cerebral metastases (unless metastases have been treated and controlled, metastases have been stable for at least 2-months post-intervention, and patient is not receiving corticosteroid treatment)
2. Certain serious illnesses or medical condition(s)
3. Has had certain other recent treatment e.g. major surgery, anticancer therapy, extended field radiation, received investigational agent, within the specified time frames prior to study drug administration
4. Has received TAS-102
5. Has unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies
6. Is a pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Every 6 weeks from the start of study treatment (Day 1, Cycle 1). Tumor assessments will be performed until radiologic progression develops or the start of new anticancer treatment.
  Tumor assessments will be performed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 every 6 weeks during study treatment, and every 8 weeks after treatment is completed. Tumor assessments will be performed from Day 1, Cycle 1 until radiologic progression develops or the start of new anticancer treatment, for up to 12 months after the last patient is randomized or until the target number of events (deaths) is met.

SECONDARY OUTCOMES:
Overall survival | Survival status will be collected at 8-week intervals until death, for up to 12 months after the first dose of study medication for the last patient randomized or until the target number of events (deaths) is met, whichever is later.
Safety monitoring including adverse events, vital signs, and laboratory assessments | Through 30 days following last administration of study medication or until initiation of new anticancer treatment
  Standard safety monitoring will be performed and adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Scagliotti, MD, Principal Investigator — University of Turin San Luigi Hospital; Kaoru Kubota, MD, PhD, Principal Investigator — Nippon Medical School Hospital Cancer Center
Locations (23):
- Germany (6):
  - Klinikum Mannheim GmbH Universitaetsklinikum, Mannheim, Baden-Wurttemberg
  - Lungenklinik Heckeshorn- HELIOS Kliniken GmbH, Berlin
  - LungenClinic Grosshansdorf, Großhansdorf
  - Klinikum Koeln-Merheim, Koplin
  - St. Hildegardis-Krankenhaus- Katholisches Klinikum Mainz, Mainz
  - LMU-Campus Innenstadt, München
- Italy (10):
  - Azienda Ospedaliero-Universitaria S. Luigi Gonzaga, Orbassano, Turin
  - IRCCS Centro di Riferimento Oncologico di Aviano, Divisione Oncologia Medica A, Aviano
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - Azienda Ospedaliera Univ. Policlinico Gaspare Rodolico, Catania
  - Azienda Ospedaliera Instituti Ospitalieri di Cremona, Cremona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera San Gerardo U.O Oncologia Medica, Monza
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - A.O.V.V. Ospedale Eugenio Morelli-Sondalo, Sondalo
- Japan (7):
  - National Cancer Center Hospital East, Chiba
  - National Kyushi Cancer Center, Fukuoka
  - Hyogo Cancer Center, Hyōgo
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - Nippon Medical School Hospital, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo

REFERENCES:
- [Derived] Scagliotti G, Nishio M, Satouchi M, Valmadre G, Niho S, Galetta D, Cortinovis D, Benedetti F, Yoshihara E, Makris L, Inoue A, Kubota K. A phase 2 randomized study of TAS-102 versus topotecan or amrubicin in patients requiring second-line chemotherapy for small cell lung cancer refractory or sensitive to frontline platinum-based chemotherapy. Lung Cancer. 2016 Oct;100:20-23. doi: 10.1016/j.lungcan.2016.06.023. Epub 2016 Jun 27. PMID 27597276